CLINICAL TRIAL: NCT02867098
Title: Pharmacokinetics and Relative Bioavailability of XmAb®5871 Administered Either Intravenously or Subcutaneously
Brief Title: XmAb5871 Bioavailability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xencor, Inc. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: XmAb5871-05
Record Dates: First submitted 2016-08-02; First posted 2016-08-15 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Healthy Volunteers
Keywords: healthy; volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1 (Experimental): Dose Level 1 XmAb5871 given SC Q14days X 3
  Interventions: Drug: XmAb5871
- Cohort 2 (Experimental): Dose Level 2 XmAb5871 given SC Q14days X 3
  Interventions: Drug: XmAb5871
- Cohort 3 (Experimental): Dose Level 3 XmAb5871 given SC Q14days X 3
  Interventions: Drug: XmAb5871
- Cohort 4 (Experimental): Dose Level 4 XmAb5871 given IV Q14days X 3
  Interventions: Drug: XmAb5871
- Cohort 5 (Experimental): Dose Level 5 XmAb5871 given SC Q7days X 3
  Interventions: Drug: XmAb5871

INTERVENTIONS:
Drug: XmAb5871

SUMMARY:
An open label comparison of concentration of the study medication administered intravenously (IV) versus subcutaneously (SC) in healthy volunteers.

DETAILED DESCRIPTION:
The study will enroll approximately 50 eligible healthy male and female subjects between the ages of 18 to 55 inclusive. There will be 5 parallel dose cohorts (Cohorts 1-5) consisting of 10 subjects in each cohort. No subject will be a member of more than 1 cohort. Subjects will receive 3 administrations of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Are adult males and females aged 18 to 55 years inclusive as of dosing (Day 1) with total body weight between 45.0 and 100.0 kg inclusive and body mass index (BMI) between 19.0 and 32.0 kg/m2 inclusive;
* Healthy as assessed by the Investigator with no clinically significant abnormality identified on medical or laboratory evaluation and no history of any clinically significant disorder, condition, or disease that would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion;

Exclusion Criteria:

* Subjects who have a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders that would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
* Subjects who are positive for drugs of abuse or alcohol on screening or admission;
* Subject is pregnant or breast feeding, or planning to become pregnant within 3 months of administration of XmAb5871.
* Subjects who have used prescription drugs (with the exception of hormonal birth control for women of child-bearing potential) within 14 days or 5 half-lives, whichever is longer, prior to dosing (Day 1), unless agreed as not clinically relevant by the Principal Investigator and Sponsor.
* Subjects who have received live vaccines ≤3 months from Day 1.
* Malignancy within 5 years (except successfully treated in situ cervical cancer, resected squamous cell or basal cell carcinoma of the skin).
* Unable or unwilling to partake in follow-up assessments or required protocol procedures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-10-21 (Actual); Study Completion 2016-10-21 (Actual)

PRIMARY OUTCOMES:
Cmax, Maximum observed serum concentration | Date of enrollment to Day 57
Tmax, Time of maximum observed serum concentration | Date of enrollment to Day 57
AUC, Area under the plasma concentration versus time curve | Date of enrollment to Day 57
CL, Clearance of drug from the body | Date of enrollment to Day 57
Vz, Volume of distribution | Date of enrollment to Day 57
F, bioavailability of a SC dose relative to an IV dose | Date of enrollment to Day 57
Number of participants with adverse events that are related to treatment | Date of enrollment to Day 57
Number of participants with severe adverse events that are related to treatment | Date of enrollment to Day 57
Number of participants with abnormal laboratory values related to treatment | Date of enrollment to Day 57
Number of participants with abnormal ECGs related to treatment | Date of enrollment to Day 57

SECONDARY OUTCOMES:
Titers of anti-XmAb5871 antibody will be assessed from time of dosing up to Day 57 | Date of enrollment to Day 57
Percent of participants positive in the assay at at least one time point | Date of enrollment to Day 57
Percent of participants with increasing titers of anti-drug antibody over time | Date of enrollment to Day 57

CONTACTS AND LOCATIONS:
Overall Officials: Esther Yoon, MD, Principal Investigator — California Clinical Trials Medical Group - PAREXEL, Early Phase Clinical Unit-Los Angeles
Locations (1):
- PAREXEL, Early Phase Clinical Unit-Los Angeles, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Kirk R, Matijevic M, Gao M, Poma A, Quinn S, Arora S, Fischer T. Pharmacokinetics, Pharmacodynamics, Bioavailability, and Immunogenicity of Obexelimab Following Subcutaneous Administration in Healthy Japanese and Non-Japanese Volunteers. Adv Ther. 2025 Feb;42(2):813-829. doi: 10.1007/s12325-024-03067-6. Epub 2024 Dec 5. PMID 39636565